CLINICAL TRIAL: NCT01867346
Title: Early Markers of Cognitive Change and Alzheimer's Disease: A Propsective Study of the Effects of Aging on Cognition and Brain Pathology
Brief Title: Early Markers of Cognitive Change and Alzheimer s Disease
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903323; 03-AG-N323
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-01-02

CONDITIONS: Alzheimer's Disease
Keywords: Cognition; Aging; Cognitive Decline; Dementia; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- The Baltimore Longitudinal Study of Aging (BLSA) is a long-term study of human aging. To see how the brain changes with age, researchers will study BLSA participants who are at least 60 years old. In particular, researchers are looking for early markers of possible Alzheimer's disease and other conditions that cause memory loss. To do so, they will give tests of memory and brain function, and stay in close contact with participants.

Objectives:

- To study cognitive changes that occur in normal aging and in people who develop memory problems.

Eligibility:

- Individuals at least 60 years of age who are participating in the BLSA.

Design:

* There are three parts to this study. These study procedures will be done under the usual BLSA guidelines.
* Participants will take paper and pencil tests. The tests measure skills such as language, attention, memory, and problem solving. They will also ask questions about emotions and feelings.
* Participants will give the name and phone number of a person who knows them well and sees them often. Researchers will ask this person to fill out questionnaires on the effects of aging on the participant. These questions will monitor the participant's memory and ability to function independently.
* Participants will have regular phone calls between study visits. These calls will help to keep their information up to date.
* Participants will continue on this study for as long as they are able to participate.

DETAILED DESCRIPTION:
Since the early 1960 s cognitive testing has been performed in conjunction with BLSA visits.

Prior to the mid-1980 s, the primary focus of these investigations was the natural history of age associated changes in memory and other cognitive functions. While a portion of the work of the Cognition Section still involves descriptive studies of cross-sectional and longitudinal effects of age on specific cognitive abilities, the cognitive testing program was refocused in the mid-1980 s to investigate early predictors of cognitive change, including risk and protective factors for cognitive impairment and Alzheimer s disease. In collaboration with Dr. Claudia Kawas, and more recently Dr. Richard O Brien of the Johns Hopkins Department of Neurology, the research program of the Cognition Section was expanded to ascertain incident cases of cognitive impairment and dementia, including home visit assessments for inactive participants. In addition, an autopsy program in collaboration with the Alzheimer s Disease Research Center (ADRC) at Johns Hopkins University was initiated. This collaboration has yielded a number of important findings including information on the incidence of Alzheimer s disease, and demonstrations that use of hormone replacement therapy in postmenopausal women and non-steroidal antiinflammatory drugs (NSAIDs) in older adults6 are associated with reductions in the risk for Alzheimer s disease in our community-dwelling BLSA participant sample.

ELIGIBILITY:
* INCLUSION CRITERIA:

All BLSA participants 60 years of age and older are included and will receive cognitive evaluations on their BLSA visits.

EXCLUSION CRITERIA:

Participants who are younger than 60 years old are excluded. Specialized testing procedures are adopted in the case of hearing or visual impairments

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2850 (Actual)
Dates: Start 2003-03-19; Primary Completion 2014-06-16 (Actual); Study Completion 2015-01-02

PRIMARY OUTCOMES:
Identifying early makers of cognitive and Alzheimer s disease | Ongoing
Characterizing risk factors which modify progression to these states | Ongoing
Cognitive changes associated with other health factors | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Alan B Zonderman, Ph.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Lindeman RD, Tobin JD, Shock NW. Association between blood pressure and the rate of decline in renal function with age. Kidney Int. 1984 Dec;26(6):861-8. doi: 10.1038/ki.1984.229. PMID 6533397
- [Background] Zonderman AB, Giambra LM, Arenberg D, Resnick SM, Costa PT Jr, Kawas CH. Changes in immediate visual memory predict cognitive impairment. Arch Clin Neuropsychol. 1995 Mar;10(2):111-23. PMID 14589733
- [Background] Troncoso JC, Martin LJ, Dal Forno G, Kawas CH. Neuropathology in controls and demented subjects from the Baltimore Longitudinal Study of Aging. Neurobiol Aging. 1996 May-Jun;17(3):365-71. doi: 10.1016/0197-4580(96)00028-0. PMID 8725897